CLINICAL TRIAL: NCT02543203
Title: Essential Oils for Enhancing of Quality of Life in Autism Spectrum Disorder (ASD)
Brief Title: Essential Oils for Enhancing QOL in ASD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jill Hollway (Other)
Collaborators: Young Living Essential Oils (Unknown)
Responsible Party: Sponsor-Investigator, Jill Hollway, Research Scientist and Assistant Professor, Research Psychiatry, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2015H0005
Record Dates: First submitted 2015-08-17; First posted 2015-09-07 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Autism Spectrum Disorder; Quality of Life; Sleep; Anxiety
Keywords: Relaxation
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A/C - Reconnect, Then Coconut Oil Comparator (Active Comparator): Participants randomized to treatment order A/C, received Reconnect for 3-months each day, morning and evening. After a washout period of one-month, they received the Coconut Oil Comparator morning and evening for 3-months.
  AM: Children received a topical application of one drop of oil to the back of the neck and 1 drop to the feet.
  PM: Children received the oil blend by the aromatic method as it was diffused throughout their bedrooms while they slept. Each bottle has an orifice that allows the oil to be expelled drop by drop the evening dose was 8-12 drops added to the diffuser.
  Interventions: Biological: Reconnect; Biological: Coconut oil Comparator
- C/A - Coconut oil Blend, Then Reconnect (Sham Comparator): Participants randomized to treatment order C/A received the Coconut Oil Comparator for 3-months each day, morning and evening. After a washout period of one-month, they received Reconnect morning and evening for 3-months.
  AM: Children received a topical application of one drop of oil to the back of the neck and 1 drop to the feet.
  PM: Children received the oil blend by the aromatic method as it was diffused throughout their bedrooms while they slept. Each bottle has an orifice that allows the oil to be expelled drop by drop the evening dose was 8-12 drops added to the diffuser.
  Interventions: Biological: Reconnect; Biological: Coconut oil Comparator

INTERVENTIONS:
Biological: Reconnect — Topical Essential Oils mixture and aromatic method
Biological: Coconut oil Comparator — Topical Essential Oils mixture and aromatic method

SUMMARY:
Essential oils (aromatic oils extracted from plant parts) are routinely used by the public and are available on the market. Investigators are conducting this study because it is unknown whether the essential oils formulations will be safe and effective for improving quality of life in children with Autism Spectrum Disorder (ASD) by helping them relax and sleep.

Children invited to participate in this study must be between 3-9 years of age and have been diagnosed with Autism Spectrum Disorder. Twenty eight children and their families will be enrolled in the study.

Participants will try two different fragrant oils in a double-blind randomized order. Each child will receive each treatment for 3 months, with a 1-month "washout" period in between during which no oil is used.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the use of two fragrant oil formulations to enhance quality of life by increasing relaxation and sleep quality in children with Autism Spectrum Disorder (ASD). Essential oils (aromatic oils extracted from plant parts) are routinely used by the public and are available on the market. Investigators are conducting this study because it is unknown whether the essential oils formulations will be safe and effective for helping children with ASD relax and sleep.

To participate in this study children must be between 3-9 years of age and have been diagnosed with Autism Spectrum Disorder. Approximately 40 children will be screened to enroll 28 children and their families in the study.

In a double-blind crossover study, participants will be randomized to treatment order. All participants will receive both fragrant oil blends. Those randomized will receive one fragrant oil blend for 3 months, with a 1-month "washout" period in between and then start the second fragrant oil blend in the last 3 months. The treatment orders are A/C and C/A.

Study participation will last for 7 months. There will be one screening visit (about 5 hours long, which can be split into 2 visits), two baseline visits (about 2 hours each), two endpoint visits (2 hours each) and 5 other clinic visits (each 45-60 minutes). Visits will take place at the OSU Nisonger Center and the OSU General Clinical Research Center.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients between 3 and 9 years of age, inclusive;
* Diagnosis of Autism Spectrum Disorder (ASD) by DSM-V;
* Mean item score of > or = 1.5 PedsQL Inventory;
* Care provider who can reliably bring subject to clinic visits and provide trustworthy ratings.

Exclusion Criteria:

* Bipolar disorder by Child & Adolescent Symptom Inventory (CASI, Gadow & Sprafkin, 1997) and clinical interview/history, or major depression accompanied by family history of bipolar disorder;
* Children with allergies to essential oils;
* Children with seizure disorder/epilepsy;
* Significant physical illness (e.g., serious cardiovascular, liver or renal pathology);
* Medications specifically given for insomnia and exogenous melatonin, which have the potential to confound study results, within the previous 2 weeks before baseline;
* Anticipated changes of doses of medication or other medical treatments or supplements;
* Weight less than 10 kg;
* Sleep Disordered Breathing (SDB) as defined by a total score of > or = 3 on the CSHQ SDB subscale and parent report;
* Nut allergies;
* Allergy to vanilla;
* A substantial trial of essential oil use within the past 6 months (i.e., consistent use for 6 weeks).

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill A Hollway, Ph.D., M.A., Principal Investigator — Ohio State University, Nisonger Center UCEDD; Eugene Arnold, M.D.,M.A., Principal Investigator — Ohio State University, Nisonger Center UCEDD
Locations (1):
- Ohio State University Nisonger Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will upload de-identified raw data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 12/30/2019
Access Criteria: Raw data in PDF archive and study report

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty subjects were screened for eligibility between between July 22nd 2015 and June 22nd 2017, at the Ohio State University's Nisonger Center.
Pre-assignment Details: Of the 40 subjects screened, 28 were randomized to treatment order. Twelve subjects did not meet the study criteria. After randomization, one subject's caregiver revealed that she could not stop melatonin treatment and another caregiver withdrew because there was a death in the family. The modified intent to treat sample included 26 participants.
Groups:
- Reconnect, Then Comparator: Participants received Reconnect each morning and evening for 3-months and then after a 1-month washout they received the comparator oil. In the morning the oil was administered topically. Participants were administered 1 drop to the back of the neck and 1 drop to the feet, to be rubbed in for 30 seconds to 1 minute.
  In the evening, before bedtime, the aromatic method was used. Caregivers diffused 8-12 drops of oil in water at night.
- Coconut Oil Comparator, Then Reconnect: Participants received the comparator oil each morning and evening for 3-months and then after a 1-month washout they received Reconnect. In the morning the oil was administered topically. Participants were administered 1 drop to the back of the neck and 1 drop to the feet, to be rubbed in for 30 seconds to 1 minute.
  In the evening, before bedtime, the aromatic method was used. Caregivers diffused 8-12 drops of oil in water at night.
Period: Overall Study
Arm/Group | Reconnect, Then Comparator | Coconut Oil Comparator, Then Reconnect
Started | 13 | 15
Completed | 7 | 10
Not Completed | 6 | 5
Not completed — Unpalatable Fragrance | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Increased Irritability | 1 | 0
Not completed — Family | 1 | 2
Not completed — Negative Behavior | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Twenty eight subjects were randomized but 2 terminated after the Baseline visit and the data analyzed was an MITT sample of 26 participant who had data for at least one other study visit from Baseline.
Groups:
- A/C (Reconnect/Comparator); C/A (Comparator/Reconnect): Topical: Apply 1 drop to the back of the neck and 1 drop to the feet. Rub in the oil for 30 seconds to 1 minute. Each bottle has an orifice that allows the oil to be expelled drop by drop. Dilution is not required, except for the most sensitive skin. Apply in the morning.
  Aromatic Method: Diffuse one diffuser-full (8-12 drops of oil in water) at night.
- Total: Total of all reporting groups
Arm/Group | A/C (Reconnect/Comparator) | C/A (Comparator/Reconnect) | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 14 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 11 | 21
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26
Children's Sleep Habits Questionnaire (CSHQ) [Mean (Full Range); unit: units on a scale 0 to 99 higher worse] | 54.25 [39 to 66] | 49.71 [33 to 72] | 51.98 [33 to 72]
Parent-rated Anxiety Scale for Autism Spectrum Disorder (PRAS-ASD) [Mean (Full Range); unit: units on a scale 0 to 75 higher worse] | 32.58 [6 to 61] | 31.71 [17 to 48] | 32.15 [6 to 61]

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Quality of Life Inventory
Description: Pediatric Quality of Life Inventory (PedsQL) (Varni, Burwinkle, & Seid, 2006). The Generic PedsQL Inventory is a caregiver-rated scale for children ages 2-12. The PedsQL Inventory for 2-4 year old children includes 21 items. The PedsQL Inventories for 5-12 year old children include 23-items. The PedsQL Inventories were designed to measure the core domains of health and their impact on the quality of life in children as outlined by the World Health Organization. The four sub-scales are Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. The summary scores include a total scale score and individual sub-scale scores. Higher scores on reversed scored items indicates better quality of life.The scores when reversed range from 0 to 100.Since there were an unequal number of items on the younger children's inventory, to be enrolled we used a cut-off of > or = 1.5 item mean on the PedsQL Inventory, which indicated poorer quality of life.
Time Frame: 28 Weeks
Population: Early terminations occurred throughout the study. Described in study flow table.
Measure: Mean (Standard Deviation); unit: Total Score
Groups:
- Subjects Received Re-Connect Then the Comparator Oil Blend: Subjects were randomized to order. Twelve subjects were randomized to Re-connect for the first 3-months, then after the one-month washout they received the coconut oil comparator during the last 3-months. The PedsQL was administered at screen, Visit 6 (at the end of the first treatment), and Visit 10 (the end of the second treatment)
- Subjects Revieved the Comparator Oil Blend and Then Re-Connnec: Subjects were randomized to treatment order. Fourteen subjects received the comparator oil blend for the first 3-months, then after the one-month washout they received Re-connect (last 3-months).The PedsQL was administered at screen, Visit 6 (at the end of the first treatment), and Visit 10 (the end of the second treatment)
Arm/Group | Subjects Received Re-Connect Then the Comparator Oil Blend | Subjects Revieved the Comparator Oil Blend and Then Re-Connnec
Number analyzed (Participants) | 12 | 14
Total Score
  Baseline Means | 45.5 (12.8) | 56.2 (5.9)
  Visit 6 Means: number analyzed (Participants) | 10 | 14
  Visit 6 Means | 61.5 (11.3) | 65.3 (8.8)
  Visit 10 Means: number analyzed (Participants) | 7 | 10
  Visit 10 Means | 64.3 (15.7) | 66.6 (5.5)

2. Secondary Outcome: Children's Sleep Habits Questionnaire
Description: Children's Sleep Habits Questionnaire (CSHQ) (Owens, Spirito, & Mcguinn, 2000). The abbreviated CSHQ is a valid measure of sleep problems with good psychometric properties. It includes 33 items and is rated retrospectively over the previous week by parents to screen for the most common sleep problems. The Abbreviated CSHQ 33 items include eight key sleep domains. The eight subscales include: (1) bedtime resistance (2) sleep onset latency, (3) sleep duration, (4) anxiety around sleep, (5) night awakenings, (6) sleep disordered breathing, (7) parasomnias and (8) morning waking/daytime sleepiness. The 33 items are summed to get a total sleep disturbance score. A total sleep disturbance score of 41 or greater for the CSHQ's 33 items has been reported to be an appropriate clinical cut-off for identifying sleep disturbance in children. Responses range from 0 to 3 with a total range of 0 to 99 for all 33 items and higher scores indicate more sleep disturbance.
Time Frame: 28 Weeks
Population: Early terminations occurred through out the study. See the Study flow table.
Measure: Mean (Standard Deviation); unit: Sleep Disturbance Total Score of 33 item
Groups:
- Subjects Received Re-Connect Then the Comparator Oil Blend: Subjects were randomized to treatment order. Twelve subjects received Re-connect for the first 3-months, then after the one-month washout they received the comparator oil blend (last 3-months).The CSHQ was administered at all visits including the Screen Visit, Visit 6 (at the end of the first treatment), and Visit 10 (the end of the second treatment).
- Subjects Received the Comparator Oil Blend and Then Re-connnec: Subjects were randomized to treatment order. Fourteen subjects received the comparator oil blend for the first 3-months, then after the one-month washout they received Re-connect (last 3-months).The CSHQ was administered at all visits including the Screen Visit, Visit 6 (at the end of the first treatment), and Visit 10 (the end of the second treatment).
Arm/Group | Subjects Received Re-Connect Then the Comparator Oil Blend | Subjects Received the Comparator Oil Blend and Then Re-connnec
Number analyzed (Participants) | 12 | 14
Sleep Disturbance Total Score of 33 item
  Baseline Means | 54.3 (7.9) | 49.7 (11.1)
  Visit 6 Means: number analyzed (Participants) | 9 | 14
  Visit 6 Means | 42.6 (6.6) | 43.1 (6.5)
  Visit 10 Means: number analyzed (Participants) | 7 | 10
  Visit 10 Means | 43.0 (6.7) | 44.5 (7.0)

3. Secondary Outcome: Parent-rated Anxiety Scale for Autism Spectrum Disorder PRAS-ASD
Description: The PRAS-ASD (Scahill et al., 2019), is a parent-rated scale used to measure anxiety in children with autism spectrum disorder. The 25 items on the PRAS-ASD each range from 0 to 3 with a possible total of 75. Higher scores indication more anxiety.
Time Frame: 28 Weeks
Population: Early terminations occurred throughout the study. See the study flow table.
Measure: Mean (Standard Deviation); unit: Total Score
Groups:
- Subjects Received Re-Connect Then the Comparator Oil Blend: Subjects were randomized to treatment order. Twelve subjects received Re-connect for the first 3-months, then after the one-month washout they received the comparator oil blend (last 3-months).The PRAS-ASD was administered at all visits including the Screen Visit, Visit 6 (at the end of the first treatment), and Visit 10 (the end of the second treatment).
- Subjects Revieved the Comparator Oil Blend and Then Re-Connnec: Subjects were randomized to treatment order. Fourteen subjects received the comparator oil blend for the first 3-months, then after the one-month washout they received the comparator oil blend (last 3-months).The PRAS-ASD was administered at all visits including the Screen Visit, Visit 6 (at the end of the first treatment), and Visit 10 (the end of the second treatment).
Arm/Group | Subjects Received Re-Connect Then the Comparator Oil Blend | Subjects Revieved the Comparator Oil Blend and Then Re-Connnec
Number analyzed (Participants) | 12 | 14
Total Score
  Baseline Means | 32.6 (15.45) | 31.7 (10.1)
  Visit 6 Means: number analyzed (Participants) | 9 | 14
  Visit 6 Means | 12.6 (11.9) | 26.4 (14.6)
  Visit 10 Means: number analyzed (Participants) | 7 | 10
  Visit 10 Means | 7.9 (5.4) | 24.0 (13.8)

4. Other Pre Specified Outcome: Developmental Disabilities - Children's Global Assessment Scale (DD=CGAS)
Description: Developmental Disabilities - Children's Global Assessment Scale (DD-CGAS) (Wagner et al., 2007). The clinician-rated DD-CGAS measures global functioning in children with developmental disorders in treatment studies. The DD-CGAS was used to characterize impairment in the following four domains: Self Care, Communication, Social Behavior, and School/Academic. In addition, this scale also includes a series of descriptive "bands" to characterize global functioning in children with pervasive developmental disorders from "extreme and pervasive impairment" through "superior functioning." Scores range fro 1 to 100 and higher scores on the DD-CGAS indicate increased independence of daily functioning.
Time Frame: 28 Weeks
Population: Early terminations occurred throughout the study. See the study flow table.
Measure: Mean (Standard Deviation); unit: Clinician Global Rating
Groups:
- Subjects Received Re-connect Then the Comparator Oil Blend: Subjects were randomized to treatment order. Twelve subjects received Re-connect for the first 3-months, then after the one-month washout they received the comparator oil blend during the last 3-months.The DDCGAS was administered at the Baseline Visit, Visit 6 (at the end of the first treatment), and Visit 10 (the end of the second treatment).
- Subjects Received the Comparator Oil Blend and Then Re-connnec: Subjects were randomized to treatment order. Fourteen subjects received the comparator oil blend for the first 3-months, then after the one-month washout they received the comparator oil blend during the last 3-months.The DDCGAS was administered at the Baseline Visit, Visit 6 (at the end of the first treatment), and Visit 10 (the end of the second treatment).
Arm/Group | Subjects Received Re-connect Then the Comparator Oil Blend | Subjects Received the Comparator Oil Blend and Then Re-connnec
Number analyzed (Participants) | 12 | 14
Clinician Global Rating
  Baseline Means | 54.8 (13.0) | 52.6 (12.7)
  Visit 6 Means: number analyzed (Participants) | 9 | 14
  Visit 6 Means | 57.9 (14.6) | 55.6 (13.5)
  Visit 10 Means: number analyzed (Participants) | 7 | 10
  Visit 10 Means | 57.4 (16.6) | 62.8 (8.8)

5. Other Pre Specified Outcome: Adverse Events
Description: Adverse Events (AEs). To minimize the risk, subjects will be systematically monitored. AEs, vital signs, including resting BP, will be evaluated at each visit throughout all phases of the study. When the treating clinician elicits an AE, it will be documented on a case report form, regardless of suspected relationship to the essential oil. For all AEs, the investigator will obtain sufficient information to determine the onset, course, and outcome of the AE. If a subject has experienced an AE, the subject may return to the site for an unscheduled visit at the PI's discretion. If any of these AEs are serious and/or unexpected, the site PI will contact the Sponsor and notify the IRB as appropriate.
  Potential AEs include sun sensitivity due to the Bergamot in the essential oil, possibly gynecomastia in pre-pubescent males due to the lavender oil in the essential oil, and skin irritation at the application site.
Time Frame: 28 Weeks
Measure: Number; unit: total number of events per condition
Groups:
- Subjects Received Re-connect Then the Comparator Oil Blend: Subjects were randomized to treatment order. Twelve subjects received Re-connect for the first 3-months, then after the one-month washout they received the comparator oil blend during the last 3-months.Adverse events were queried by the study physician at all study visits. Safety population included all participants who received one dose of study IP.
- Subjects Received the Comparator Oil Blend and Then RE-connect: Subjects were randomized to treatment order. Fourteen subjects received the comparator oil blend for the first 3-months, then after the one-month washout they received Re-connect during the last 3-months. Adverse events were queried by the study physician at all study visits.
Arm/Group | Subjects Received Re-connect Then the Comparator Oil Blend | Subjects Received the Comparator Oil Blend and Then RE-connect
Number analyzed (Participants) | 12 | 14
total number of events per condition
  Visit 6 | 27 | 35
  Visit 10 | 34 | 18

ADVERSE EVENTS:
Time Frame: Participants are systematically monitored for adverse events by study physicians (at all 10 visits). Vital signs, including resting BP, were evaluated at every visit as well.
Description: According to all laboratory reports and physician review of adverse events potentially related to oil blend administration, there are no clinically significant abnormal values or adverse events. Recorded adverse events related to study treatment include minor events such as hyperactivity and intolerance to oil smell
Groups:
- Reconnect: Subjects were randomized to treatment order in a cross-over study design. The adverse events noted below were recorded from subjects in the Reconnect group.
- Coconut Oil Blend (Comparator): Subjects were randomized to treatment order in a cross-over study design. The adverse events noted below were recorded from subjects in the coconut oil comparator group.
Arm/Group | Reconnect | Coconut Oil Blend (Comparator)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 24/24 | 23/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reconnect (N=24) | Coconut Oil Blend (Comparator) (N=23)
URI (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) — Upper respiratory infection
Increased Irritability (Psychiatric disorders) | 4 (4) | 1 (1) — Increased Irritability
Streptococcal pharyngitis, (Infections and infestations) | 3 (3) | 1 (1) — Streptococcal pharyngitis
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6) — Vomiting
Enuresis (Renal and urinary disorders) | 2 (2) | 2 (2) — Enuresis
Environmental Allergy (Immune system disorders) | 2 (2) | 3 (3) — Allergy
Tussis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) — Tussis or cough
Fever (Infections and infestations) | 2 (2) | 2 (2) — Fever
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 3 (3) — Gastroenteritis
Gastrointestinal upset (Gastrointestinal disorders) | 2 (2) | 0 (0) — Gastrointestinal upset
Increased Self Injury (Psychiatric disorders) | 1 (1) | 2 (2) — Increased Self Injury (biting self)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 2 (2) — Otitis media
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — Rhinorrhea
Sleep disturbance (Psychiatric disorders) | 0 (0) | 2 (2) — Sleep disturbance
Viral exanthem (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Exanthem rash or eruption on the skin due to virus
Increase of verbal stemming (Psychiatric disorders) | 0 (0) | 3 (3) — Increase in verbal stemming (squealing)
Adverse reaction to noxious oil smell (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Noxious oil smell

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT02543203/Prot_SAP_000.pdf